CLINICAL TRIAL: NCT05838781
Title: DeteCtiON and Stroke PreventIon by MoDEl ScRreenING for Atrial Fibrillation
Acronym: CONSIDERING-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Region Halland (Other); Halmstad University (Other); Karolinska Institutet (Other); Pfizer (Industry); Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Johan Engdahl, MD, Associate Professor, Senior consultant, Karolinska Institutet, Bristol-Myers Squibb
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: CV185-837
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Mass Screening
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Intervention Model Description: Siteless, randomized, 2x2 factorial design, superiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- General/control (No Intervention): Standard of care.
- General/intervention (Experimental): Standard of care plus 14-days continuous ECG monitoring using an ECG patch.
  Interventions: Diagnostic Test: 14-days continuous ECG monitoring
- Risk prediction model/control (Experimental): Standard of care.
  Interventions: Diagnostic Test: Risk prediction model
- Risk prediction model/intervention (Experimental): Standard of care plus 14-days continuous ECG monitoring using an ECG patch.
  Interventions: Diagnostic Test: Risk prediction model; Diagnostic Test: 14-days continuous ECG monitoring

INTERVENTIONS:
Diagnostic Test: Risk prediction model — A risk prediction model (RPM) based on logistic regression. The RPM uses 13 variables accessible in healthcare registers to identify individuals with high future risk for developing AF. ICD-10 codes will be used.
  Arms: Risk prediction model/control; Risk prediction model/intervention
Diagnostic Test: 14-days continuous ECG monitoring — 14-days continuous ECG monitoring with an ECG patch.
  Arms: General/intervention; Risk prediction model/intervention

SUMMARY:
Atrial fibrillation (AF) is the most common clinical arrhythmia and the prevalence increases with age. AF increases the risk of ischaemic stroke fivefold and accounts for almost one-third of all strokes. As AF is often asymptomatic there are many undetected cases. It is important to find patients with AF and additional risk factors for stroke in order to initiate oral anticoagulation treatment, which can reduce the risk of an ischaemic stroke by 60-70%. Screening is recommended in European guidelines, however the most suitable population and the most suitable device for AF detection remain to be defined.

The main objective of this study is to test the hypothesis that AF screening with 14-days continuous ECG monitoring in high-risk individuals identified with a risk prediction model is more effective than routine care in identifying patients with undetected AF.

Effectively detecting AF among patients with risk factors for ischaemic stroke has the potential to decrease mortality and morbidity, stroke burden and costs for the society as a whole.

DETAILED DESCRIPTION:
Objective(s): To compare the yield of atrial fibrillation (AF) using 14-days continuous ECG in a population aged ≥ 65 years with an increased risk for AF incidence according to the risk prediction model compared with standard of care in Region Halland.

Study Population: Residents in Region Halland age 65 and above.

Data Collection Methods: Electronic Health Records from Region Halland and 14-days continuous ECG recording using an ECG patch.

Study design:

Step 1:

To calibrate the BMS/Pfizer risk prediction model (RPM), we will extract two cohorts retrospectively: the AF cohort with an AF diagnosis (patients with a record of incident AF diagnosis between January 1, 2016, and December 31, 2019 as an observation period), and the control cohort without any AF diagnosis in their history. We will include patients ≥45 years of age at index date, which is the first date of an AF diagnosis recorded in the observation period and a random pseudo index date during the observation period for the control group, to follow the original study. Specifically, we are looking to calibrate the intercept (α) for the logistic regression where we already have the 13 odd ratios for the 13 risk factors from the original study. Then in the next step for the prospective study, applying the RPM on the RPM cohort, the at-risk group will be extracted for randomization step, using the recommended cut-off value.

Step 2:

The population in Region Halland aged 65 years and above and free from AF will be randomized into two halves, creating a general cohort and an RPM cohort. In the general cohort, 1480 individuals will be further randomized into two arms, general/control and general/intervention. In the RPM cohort, the risk of incident AF will be calculated according to the Pfizer/BMS RPM. Those with a predicted risk for incident AF above a pre-specified threshold will then be randomly extracted into two arms, RPM/control and RPM/intervention (figure 1).

Those randomized to the two intervention arms (general/intervention and RPM/intervention, n=740 each) will be invited to an AF screening intervention of 14-days continuous ECG using a patch device. Those randomized to the control groups (general/control and RPM/control, n=740 each) will not receive any information or intervention.

The primary endpoint will be the difference in yield of newly diagnosed AF between the RPM/intervention and the general/control arms, where the latter will represent standard of care. Participants with newly diagnosed AF in the intervention arms will be offered consultation aiming at AF work-up and initiation of oral anticoagulation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Alive residents in the Halland region aged 65 or older without a recorded diagnosis of AF

Exclusion Criteria:

* Known atrial fibrillation
* Death
* No longer resident in Region Halland
* Pacemaker, implantable cardioverter defibrillator or insertable monitor
* Dementia
* Other indication for OAC treatment (such as VTE, mechanical heart valve replacement, VTE prophylaxis post surgery, mitral stenosis, left side intracardial thrombus)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2112 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Incident AF | 14 days
  1. Incident AF on ECG screening (intervention arms) defined as at least one episode of AF or atrial flutter with a duration of at least 30 seconds on ambulatory ECG recording.
  2. Incident AF registered in the Electronic Health Record during follow-up (all four arms).

SECONDARY OUTCOMES:
Yield newly diagnosed AF: RPM/ intervention arm versus RPM/ control arm | 14 days
  To compare the yield of newly diagnosed AF using 14-days continuous ECG in a population aged ≥ 65 years with an increased risk for AF incidence according to the RPM compared with a population with increased risk according to the RPM without intervention.
Yield newly diagnosed AF: general/ intervention arm versus RPM/ control arm | 14 days
  To compare the yield of newly diagnosed AF using 14-days continuous ECG in a general population aged ≥ 65 years compared with a population with increased risk according to the RPM without intervention.
Yield newly diagnosed AF: general/ intervention arm versus general/ control arm | 14 days
  To compare the yield of newly diagnosed AF using 14-days continuous ECG in a general population aged ≥ 65 years compared with a general population without intervention.

OTHER OUTCOMES:
Proportion of patients starting oral anticoagulation treatment | 18 months
  Proportion of patients with AF and treatment with anticoagulation in control and interventions arms in the general and RPM cohorts, respectively, during a 6-, 12- and 18-months period?
Feasibility of self-application of ECG patch | 14 days
  To study uptake and feasibility of self-application of ECG patch.
AF yield during the first 24 and 48 hours | 48 hours
  Proportion of patients diagnosed with AF within the first 24 and 48 hours of ECG patch recording.
Cost-effective analysis | 14 days
  Cost-effectiveness analysis of the risk prediction model together with the ECG patch compared to standard care. The possibility to increase survival as a consequence of avoiding AF-related events will then be compared to increased screening costs as well as cost of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Engdahl, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet Danderyd University Hospital, Stockholm, Outside US
  - Halland Hospital Varberg, Varberg, Outside US

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Etminani F, Sandgren E, Holm J, Magnusson P, Modica A, Moberg K, Davidsson T, Stalpe L, Kiflemariam S, Younan N, Parikh P, Wadhwa M, Sundin A, Engdahl J. Randomised, siteless study to compare systematic atrial fibrillation screening using enrichment by a risk prediction model with standard care in a Swedish population aged >/= 65 years: CONSIDERING-AF study design. BMJ Open. 2024 Jan 12;14(1):e080639. doi: 10.1136/bmjopen-2023-080639. PMID 38216189